CLINICAL TRIAL: NCT00454298
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Regimen, Parallel-Group Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AGG-523 Administered Orally to Subjects With Severe Osteoarthritis
Brief Title: Study Evaluating AGG-523 in Subjects With Severe Osteoarthritis Requiring Total Knee Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3189A1-106
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
Keywords: Severe Osteoarthritis; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Active Comparator): AGG-523 1800 mg QD PO (12 capsules) for 28 days
  Interventions: Drug: AGG-523 (Aggrecanase Inhibitor)
- B (Active Comparator): AGG-523 900 mg BID PO (12 capsules) for 28 days
  Interventions: Drug: AGG-523 (Aggrecanase Inhibitor)
- C (Placebo Comparator): Placebo QD PO (12 capsules) for 28 days
  Interventions: Drug: AGG-523 (Aggrecanase Inhibitor)
- D (Placebo Comparator): Placebo BID PO (12 capsules) for 28 days
  Interventions: Drug: AGG-523 (Aggrecanase Inhibitor)

INTERVENTIONS:
Drug: AGG-523 (Aggrecanase Inhibitor)

SUMMARY:
The main purpose of the study is to find out if, after 4 weeks of dosing, signs of the investigational drug AGG-523, or its effects, can be measured in urine, blood, or the knee joint. A secondary purpose is to evaluate the safety of taking the drug either once a day or twice a day for 4 weeks.

DETAILED DESCRIPTION:
This is a multicenter study of 2 dosing regimens of AGG-523, an investigational aggrecanase inhibitor that is taken orally. Potential study subjects are those with severe Osteoarthritis (OA) of the knee who are scheduled to undergo total joint replacement surgery.

Study subjects will be randomly assigned to 1 of 2 dosing regimens (once-daily or twice-daily dosing) of either 1800 mg AGG-523 or placebo, which will be taken during the 4-week period before having the total knee replacement. The treatments will be assigned using a 4:1 ratio of active to placebo treatment, which means that more subjects will receive the active treatment than the placebo (see below).

* AGG-523 1800 mg once a day (32 subjects)
* AGG-523 900 mg twice a day (32 subjects)
* Placebo once a day (8 subjects)
* Placebo twice a day (8 subjects)

Study subjects will have weekly evaluations as outpatients during the 4-week dosing period. The purpose of these evaluations is to monitor for potential complications, ensure compliance with taking the study drug, ask about the use of other medications, and, when necessary, replenish the supply of study drug. These assessments may be conducted by telephone, as a home visit, or by having the subject travel to the clinic for an outpatient office visit. A final (in person) visit will happen 2 weeks after having total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, men or women, at least 55 years old
* Osteoarthritis of the knee requiring total knee replacement surgery

Exclusion Criteria:

* Other types of arthritis, like rheumatoid arthritis
* Recent major surgery (in past 3 months)
* Recent knee injections (in past 6 months)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Using parts of the knee joint and the surrounding fluid that is taken out at the time of knee replacement, measure 1) the activity of aggrecansase (an enzyme that breaks down cartilage) and 2) the amount of study drug using lab tests. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Montior, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- United States (4):
  - Boston, Massachusetts
  - Newton, Massachusetts
  - Winchester, Massachusetts
  - Worcester, Massachusetts